CLINICAL TRIAL: NCT07028554
Title: Post-Market Clinical Follow-Up Study Plan for Cartridges of Disposable Endoscopic Linear Cutting Staplers
Status: Recruiting | Type: Observational
Sponsor: Suzhou Kerui Medical Technology Co., Ltd (Other)
Responsible Party: Sponsor
Other Study IDs: WEKD-QS-PMCF
Record Dates: First submitted 2025-06-03; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: the Transection of Tissues; the Resection of Tissues; the Creation of Anastomoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cartridges of Disposable Endoscopic Linear Cutting Staplers: Investigational devices are Cartridges of Disposable Endoscopic Linear Cutting Staplers, Disposable Powered Endoscopic Linear Cutting Staplers and Disposable Endoscopic Linear Cutting Staplers manufactured by Ningbo Verykind Medical Device Co., Ltd.
  Interventions: Device: Cartridges of Disposable Endoscopic Linear Cutting Staplers, Disposable Powered

INTERVENTIONS:
Device: Cartridges of Disposable Endoscopic Linear Cutting Staplers, Disposable Powered — Investigational devices encompassing all models of the Cartridges for Disposable Endoscopic Linear Cutting Staplers, as well as Staplers utilized in conjunction with the Cartridges specified in the Study Plan (Plan number: WEKD-QS-PMCF).

SUMMARY:
Cartridges of Disposable Endoscopic Linear Cutting Staplers, Disposable Powered Endoscopic Linear Cutting Staplers and Disposable Endoscopic Linear Cutting Staplers manufactured by Ningbo Verykind Medical Device Co., Ltd. have marketed in many countries or area for many years. The investigational devices are intended for transection, resection, and/or creation of anastomoses. The instruments have application in multiple open or minimally invasive general, gynecologic, urologic and thoracic surgical procedures.

In order to confirm the safety and performance of the products, as well as the continued safety and clinical performance of the implant (the staple) during the clinical follow-up period, monitor the identified side-effects, contraindications and identify previously unknown side-effects, and ensure the continued acceptability of the benefit-risk ratio, Investigators proactively collect and evaluate clinical data from different regions, including of Italy, Brazil and Chile, where the device has been marketed, and conduct PMCF studies.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years old, gender unlimited;
2. The surgery type shall be open or endoscopic surgery;
3. The departments of surgical procedures: general, gynecologic, urologic and thoracic surgical procedures;
4. Investigational devices listed in this PMCF plan must be used during surgical procedures.

Exclusion Criteria:

1. Patients with surgical contraindications to the product, e.g. use the instruments on large arteries, on ischemic or necrotic tissue, use the device on tissues with a compression thickness out of the device range;
2. Concomitant with similar devices (staplers/reloads/cartridges, etc.) for resection, transection and anastomosis of surgical organ or tissues;
3. The operation record is incomplete, and the information related to the main indicators cannot be extracted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cartridges of Disposable Endoscopic Linear Cutting Staplers are intended for transection, resection, and/or creation of anastomoses. The instruments are applied in multiple open or minimally invasive general, gynecologic, urologic and thoracic surgical procedures. They must be used in combination with Disposable Powered Endoscopic Linear Cutting Staplers or Disposable Endoscopic Linear Cutting Staplers manufactured by the Company.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Anastomosis success rate | The investigation sites will be collected from January 2023 to June 2024.
  According to surgical records and inpatient medical records, no reoperation in situ is defined as successful anastomosis.

SECONDARY OUTCOMES:
Anastomotic bleeding rate | The incidence of anastomotic bleeding during day of operation and 6 months after operation was recorded.
Anastomotic leakage rate | The incidence of leakage during day of operation and 6 months after operation was recorded.
Anastomotic stenosis rate | The incidence of anastomotic stenosis during day of operation and 6 months after operation was recorded.

OTHER OUTCOMES:
Surgical time | The investigation sites will be collected from January 2023 to June 2024.
Intraoperative bleeding | The investigation sites will be collected from January 2023 to June 2024.
Intraoperative conversion (due to device reasons) | The investigation sites will be collected from January 2023 to June 2024.
Length of hospitalization | The investigation sites will be collected from January 2023 to June 2024.

CONTACTS AND LOCATIONS:
Locations (1):
- Cartridges of Disposable Endoscopic Linear Cutting Staplers, Ningbo, Zhejiang, Chile

IPD SHARING:
Plan to Share IPD: No